CLINICAL TRIAL: NCT02866838
Title: Treatment of Intracerebral Hemorrhage in Patients on Non-vitamin K Antagonist Oral Anticoagulants (NOAC) With Tranexamic Acid
Brief Title: Treatment of Intracerebral Hemorrhage in Patients on Non-vitamin K Antagonist
Acronym: TICH-NOAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BASEC 2016-01251
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Tranexamic acid; NOAC; Direct Oral Anticoagulant (DOAC); Direct oral anticoagulants; Non-Vitamin K antagonist oral anticoagulants
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Intravenous tranexamic acid: 1g loading dose given as 100 mls infusion over 10 minutes, followed by another 1g in 250 mls infused over 8 hours.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Saline 0.9% given in identical dosage as experimental
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Tranexamic acid — intravenous
  Other Names: Cyklokapron
  Arms: Tranexamic acid
Drug: Saline 0.9% — intravenous
  Arms: Placebo

SUMMARY:
Novel, non-vitamin K antagonist oral anticoagulants (NOAC) target selected players in the coagulation cascade as the direct thrombin inhibitor dabigatran and the factor Xa-inhibitors apixaban and rivaroxaban. Intracerebral hemorrhage (ICH) is the most feared complication of NOAC treatment (NOAC-ICH).

Outcome of NOAC-ICH can be devastating and is a major cause of death and disability. There is no proven treatment for NOAC-ICH. Hematoma expansion (HE) is associated with unfavorable outcome. Tranexamic acid (TA) is an anti-fibrinolytic drug that is used in a number of bleeding conditions other than ICH.

ELIGIBILITY:
Inclusion Criteria:

* Acute intracerebral hemorrhage (symptom onset <12h)
* Prior treatment with a novel direct oral anticoagulant (apixaban, dabigatran, edoxaban or rivaroxaban; last intake <48hours or proven NOAC activity by relevant coagulation assays)
* Age >18 years, No upper age limit
* Informed consent has been received in accordance to local ethics committee requirements

Exclusion Criteria:

* Severe pre-morbid disability (modified Rankin scale >4)
* Anticoagulation with Vitamin K antagonists (VKA) (recent intake)
* Secondary intracerebral hemorrhage (e.g. arteriovenous malformation (AVM), tumor, trauma) Note it is not necessary for investigators to exclude underlying structural abnormality prior to enrolment, but where an underlying structural abnormality is already known, these patients should not be recruited.
* Glasgow coma scale <5
* pregnancy
* Planned neurosurgical hematoma evacuation within 24 hours (before follow-up imaging)
* Pulmonary embolism/deep vein thrombosis within the last 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Hematoma expansion | up to 27 hours
  Change in ICH-volume between baseline CT and follow-up-CT at 24 ± 3 hours of 33% relative or 6ml absolute increase

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) 0-4 at month 3; | 3 months
mRS 0-3 at month 3; | 3 months
Categorical shift in mRS at month 3 | 3 months
mortality due to any cause at month 3 | 3 months
In-hospital mortality | baseline until discharge from hospital (stay at hospital lasts on an average of 10 days)
Absolute ICH growth volume by 24 ± 3 hours, adjusted for baseline ICH volume | up to 27 hours
Symptomatic HE defined as HE and additionally a neurological deterioration of NIHSS >4 points or Glasgow Coma Scale (GCS) >2 points | up to 27 hours
number of major thromboembolic events (myocardial infarction, ischemic stroke, pulmonary embolism - safety endpoints) | 3 months
number of neurosurgical interventions (including craniectomy, external ventricular drain (EVD), hematoma evacuation) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lyrer, MD, Study Chair — Stroke Center and Neurology, University Hospital Basel; Stefan Engelter, MD, Study Chair — Stroke Center and Neurology, University Hospital Basel
Locations (1):
- Stroke Center, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Polymeris AA, Karwacki GM, Siepen BM, Schaedelin S, Tsakiris DA, Stippich C, Guzman R, Nickel CH, Sprigg N, Kagi G, Vehoff J, Barinka F, Thilemann S, Maurer M, Wagner B, Traenka C, Gensicke H, De Marchis GM, Bonati LH, Fischer U, Z'Graggen WJ, Nedeltchev K, Wegener S, Baumgartner P, Engelter ST, Seiffge DJ, Peters N, Lyrer PA; TICH-NOAC Investigators. Tranexamic Acid for Intracerebral Hemorrhage in Patients on Non-Vitamin K Antagonist Oral Anticoagulants (TICH-NOAC): A Multicenter, Randomized, Placebo-Controlled, Phase 2 Trial. Stroke. 2023 Sep;54(9):2223-2234. doi: 10.1161/STROKEAHA.123.042866. Epub 2023 Jul 19. PMID 37466000

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT02866838/Prot_SAP_000.pdf